CLINICAL TRIAL: NCT06390007
Title: The Efficacy of Acupuncture in the Management of Postoperative Pain in the Pediatric Intensive Care Unit at Cipto Mangunkusumo Hospital
Brief Title: The Efficacy of Acupuncture in the Management of Postoperative Pain in the Pediatric Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Irene Yuniar, Sp.A(K), Lecturer of Indonesia University, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24916
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Pain, Postoperative; Pediatric Disorder; Acupuncture; Acupuncture, Ear; Pediatric Intensive Care Unit
Keywords: Acupuncture; Postoperative pain; Pediatric Intensive Care Unit; Press needle; Pain therapy
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): In the control group, standard analgesic therapy will be administered by the attending physician, and a sham press needle (a patch resembling a press needle without a needle) will be applied.
  Interventions: Device: Sham press needle
- Intervention group (Experimental): In the experimental group, standard analgesic therapy will be administered and press needle acupuncture will be applied at acupuncture points.
  Interventions: Device: Press needle acupuncture

INTERVENTIONS:
Device: Sham press needle — The plester used is a round plaster that resembles the shape of an acupuncture press needle.
  Other Names: plesterin
  Arms: Control group
Device: Press needle acupuncture — Press needle acupuncture is a modality of acupuncture using tiny and very thin needles.
  Arms: Intervention group

SUMMARY:
Pain is an unpleasant sensory and emotional experience resulting from tissue damage. Pain management is typically conducted according to the World Health Organization (WHO) pain management ladder. Analgesics administered to pediatric patients vary in dosage and type, but these analgesics often have significant side effects. The acupuncture technique using press needles is a non-pharmacological pain therapy modality that has been studied for its ability to reduce the use of analgesic drugs, thereby potentially decreasing side effects associated with analgesic use.

The study was conducted using a randomized controlled trial (RCT) design involving 70 pediatric postoperative patients aged 1-18 years who were admitted to the Pediatric Intensive Care Unit at Cipto Mangunkusumo Hospital. Subjects were divided into two groups: a control group and an experimental group. The control group received standard analgesic therapy and sham press needle application (a patch resembling a press needle without a needle), while the experimental group received standard analgesic therapy and press needle application at acupuncture points after the patient had been in the Pediatric Intensive Care Unit for 24 hours. Pain scale monitoring was conducted at 1, 6, 24, 48, and 72 hours using the Face, Legs, Activity, Cry, and Consolability (FLACC) scale for children aged 1-8 years, and the Numeric Rating Scale (NRS) for children over 8 years old.

This study hypothesizes that the acupuncture technique using press needles can reduce the pain scale in pediatric postoperative patients, leading to a decrease in the use of analgesics and a reduction in side effects associated with analgesic use.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric postoperative patients admitted to the Pediatric Intensive Care Unit at Cipto Mangunkusumo Hospital
* Aged between 1 and 18 years
* Patients with a platelet count greater than 20,000/mL
* Patients undergoing elective surgery
* Willingness to participate in the study

Exclusion Criteria:

* Patients with a local infection at the puncture site
* Patients with anatomical abnormalities of the outer ear
* Failure to complete the acupuncture therapy
* Patients with chronic illnesses who have previously received analgesic therapy

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-03-22 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Face, Legs, Activity, Cry, and Consolability (FLACC) pain scale | Pain scale monitoring will be conducted at 1 hour; 6 hours; 24 hours; 48 hours; and 72 hours after the application of sham press needle / press needle acupuncture
  The Face, Legs, Activity, Cry, and Consolability (FLACC) pain scale for children aged 1 to 8 years is used to assess pain levels
Numeric Rating Scale (NRS) pain scale | Pain scale monitoring will be conducted at 1 hour; 6 hours; 24 hours; 48 hours; and 72 hours after the application of sham press needle / press needle acupuncture
  The Numeric Rating Scale (NRS) is used to assess pain levels in children over the age of 8.
Behavioral Pain Scale (BPS) | Pain scale monitoring will be conducted at 1 hour; 6 hours; 24 hours; 48 hours; and 72 hours after the application of sham press needle / press needle acupuncture
  The Behavioral Pain Scale (BPS) with a range of 3 to 12 for patients on ventilators.

CONTACTS AND LOCATIONS:
Locations (1):
- RSUPN Dr. Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No